CLINICAL TRIAL: NCT03766022
Title: Effect of Heavy Smoking on Hard and Soft Tissue Parameters Prospective Controlled Clinical Trial
Brief Title: Effect of Heavy Smoking on Hard and Soft Tissue Parameters Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CTIL-0418-18-RMB
Record Dates: First submitted 2018-11-20; First posted 2018-12-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Dental Implants,Peri-implantitis,Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heavy smoker patients (Experimental): Marginal bone changes after 1 year after implant installation using Neo dental implant Alpha Bio Tec. Ltd.
  Interventions: Device: Neo dental implant Alpha Bio Tec. Ltd.
- non Smokers patients (Active Comparator): Marginal bone changes after 1 year after implant installation using Neo dental implant Alpha Bio Tec. Ltd.
  Interventions: Device: Neo dental implant Alpha Bio Tec. Ltd.

INTERVENTIONS:
Device: Neo dental implant Alpha Bio Tec. Ltd. — Neo dental implant is used to restore missing teeth

SUMMARY:
The Aim of this study randomized prospective clinical trial is to examine and compare periimplant tissue changes between heavy smokers and non-smokers at 12 months post loading using the alpha Bio Neo standard diameter implants with conical abutment.

DETAILED DESCRIPTION:
Peri-implant marginal bone level is one of the most important references criteria to monitor peri-implant health.A radiographically measured marginal bone loss of up to 1.5 mm during the first year of loading, followed by a marginal bone loss of up to 0.2 mm for each succeeding year, is an acceptable criterion to determine implant success.

Smoking has been implicated in many adverse systemic outcomes, including tooth loss, alveolar bone loss and dental implant failure.

Platform switching, also known as platform shifting, is whenever an abutment is used that is smaller in diameter than the implant platform. Platform switching can help prevent crestal bone loss.

The hypothesis of the present study is that the use of conical abutment might reduce marginal bone loss around dental implants in both smokers and non-smokers alike.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 - 85 years.
2. Written informed consent.
3. In need for a dental implant Adequate alveolar bone Intended to be restored with individual crowns.
4. Heavy smokers (20 Cig/d > 5years) or non / former smokers (> 5 years since cessation).

Exclusion Criteria:

1. Active periodontal disease.
2. Systemic condition and medication that may affect soft and hard tissue.
3. healing Parafunctional occlusal scheme and habits.
4. Pregnancy or intention to become pregnant in the following twelve months.
5. Patient not willing or able to meet the study schedule.
6. Patient in need for simultaneous bone graft or GBR using a membrane barrier.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | 6 months and 18 months after implantation.
  Standardized periapical radiographs will be used to assess changes in radiographic bone height.

SECONDARY OUTCOMES:
Implants probing depth (IPD) | 4 months, 6 months and 16 months after implantation
  will be measured by inserting a probe to the gingival pocket at six sites around implant
Bleeding on probing | 4 months, 6 months and 16 months after implantation
  will be measured by inserting a probe to the gingival pocket at six sites around each implant: Dichotomic measurments: Yes/No
Labial gingival recession | 4 months, 6 months and 16 months after implantation
  will be measured using the incisal edge. occlusal plan as a fixed reference point.

OTHER OUTCOMES:
Implant stability | Immediatly after implant installation (day 0) and 4 months after implantation
  Osstel measurements

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Zigdon, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Hospital, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No